CLINICAL TRIAL: NCT03540810
Title: Hydroxychloroquine Versus Placebo: Impact on Thrombotic Relapse in Primary Antiphospholipid Syndrome
Acronym: PAPIRUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-004416-19
Record Dates: First submitted 2018-04-27; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Primary Antiphospholipid Syndrome
Keywords: antiphospholipid syndrome; thrombosis; hydroxychloroquine
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombosis | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): All patients randomised in this arm will receive hydroxychloroquine with their usual treatment, which is antivitamin K anticoagulants
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): All patients randomised in this arm will receive a placebo with their usual treatment, which is antivitamin K anticoagulants
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — The patients will additionally receive this drug with their usual treatment to evaluate its efficiency to prevent new thrombotic events in primary antiphospholipid syndrome patients
  Other Names: HCQ
  Arms: Hydroxychloroquine
Drug: Placebo — The patients will receive placebo with their usual treatment
  Arms: Placebo

SUMMARY:
Antiphospholipid syndrome (APS) combines thrombotic (venous and/or arterial) and/or obstetrical manifestations, along with biological anomalies related to the presence of antiphospholipid antibodies. Despite actual treatment recommended by international guidelines, the relapse rate in APS is high and survival is 65% at 15 years. Hydroxychloroquine has demonstrated its efficacy and benefits in the treatment of Systemic Lupus Erythematosus, but there is no current consensus concerning the efficacy of this treatment in the secondary prevention of thrombotic events in primary APS, even though several in vitro experimental and animal model data, along with several clinical studies have suggested a beneficial effect of this drug in this indication. Considering the prevalence of primary APS in the general population and of the number of clinical events observed in patients with primary APS and receiving conventional treatment with vitamin K anticoagulants (VKA), the consortium expects a minimum clinically relevant difference of 70%. Considering a prevalence of thrombotic events for the entire studied primary APS population of 10% at 2 years, the consortium expects a 70% decrease in thrombotic events under Hydroxychloroquine treatment administered in addition to VKA treatment in primary APS, i.e. a 3% prevalence in the Hydroxychloroquine group at 2 years. The consortium proposes a drug trial, phase III, national multicentric, comparative, randomized, superiority, double-blind, controlled with 2 compared groups (Hydroxychloroquine versus placebo) study. The enrolment period will be 24 months.

The main aim of this trial is to comparatively assess at 24 months the number of new thrombotic events (venous and arterial) in primary antiphospholipid syndrome in patients treated with VKA plus Hydroxychloroquine versus VKA plus placebo, in a multicentre, prospective randomized, double-blind, versus placebo study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Presence of a primary antiphospholipid syndrome with previous venous/arterial thrombosis and which needs a treatment with VKA
* Patients with a signed commitment

Exclusion Criteria:

* Secondary APS
* Ocular diseases :

  * retinal disease contraindicating the prescription of hydroxychloroquine
  * cataract
  * monophtalmic
* Past history of intolerance or allergy to hydroxychloroquine
* Known deficit in G6PDase
* Hemolytic anemia
* Porphyria
* Chronic hepatic disease
* Severe renal failure (creatinin clearence <30ml/min)
* Chronic alcoholism
* Patient with QT interval >440 ms on the ECG
* Concomitant treatment with drugs raising the QT interval
* Epilepsy
* Pregnant or breastfeeding women
* Women refusing an effective contraception
* Active cancer or malignant hemopathy
* Psychiatric disease unabling the compliance to treatment
* Unaffiliated person or not beneficiary of a social security system
* Concomitant participation at a biomedical trial able to interfere with the actual trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of thrombotic events in each arm after 24 months of treatment | 24 month
  The number of thrombotic events will be compared in the two arms of the study. The events which will be considered are deep venous thrombosis, superficial venous thrombosis, lung embolism, stroke, myocardial infarction as assessed by at least one diagnostic tests such as: doppler echography, lung scintigraphy, lung CT scan, cerebral CT scan, cerebral MRI, myocardial scintigraphy, coronarography.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE | 24 month
  The number of participants with treatment-related adverse events as assessed by CTCAE will be compared in the two arms of the study
Number of hospitalizations days related to thrombotic event | 24 month
  The number of hospitalizations days, related to thrombotic event in each arm after 24 months of treatment
Number of work incapacity days related to thrombotic event | 24 month
  The number of work incapacity days, related to thrombotic event in each arm after 24 months of treatment
The specific biological markers of thrombosis in APS such as type and number of antiphospholipid antibodies, complement, antinuclear antibodies, thrombocytosis | 24 month
  The specific biological markers of thrombosis in APS such as type and number of antiphospholipid antibodies, complement, antinuclear antibodies, thrombocytosis in each arm
Assess compliance to VKA | 24 month
  The different recorded values of blood INR all along the study
Assess Assess compliance to HCQ | 24 month
  The values of blood Hydroxychloroquine measured at the end of the 24 months of treatment
The vascular arterial rigidity measured by doppler echography | 24 month
  The vascular arterial rigidity measured by doppler echography will be compared between the two arms of the study at inclusion in the study and after 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Belizna, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- University Hospital Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No